CLINICAL TRIAL: NCT07267481
Title: Efficacy of Switching Participants Treated With Xiidra to TRYPTYR
Brief Title: Switching From Xiidra to TRYPTYR
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Southern College of Optometry (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00006763-Xiidra
Record Dates: First submitted 2025-11-25; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Dry Eye; Dry Eyes Chronic; Dry Eye Syndromes; Eye Diseases
MeSH Terms: conditions — Dry Eye Syndromes; Eye Diseases

STUDY DESIGN:
Intervention Model Description: This prospective, single-masked (participant), single-armed, study will determine how participants who are being treated with Xiidra respond to acoltremon 0.003%
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- acoltremon (Experimental): Switching to acoltremon 0.003% will significantly improve the signs and symptoms of participants who were being treated with Xiidra at 28 days post-treatment compared to baseline.
  Interventions: Drug: acoltremon 0.003%

INTERVENTIONS:
Drug: acoltremon 0.003% — Switching to acoltremon 0.003% will significantly improve the signs and symptoms of participants who were being treated with Xiidra at 28 days post-treatment compared to baseline.

SUMMARY:
To determine the efficacy of switching participants who are being treated with Xiidra to acoltremon 0.003%.

Hypothesis: Switching to acoltremon 0.003% will greatly improve the signs and symptoms of participants who were being treated with Xiidra at 28 days post-treatment compared to baseline.

DETAILED DESCRIPTION:
This prospective, single-masked (participant), single-armed, study will determine how participants who are being treated with Xiidra respond to acoltremon 0.003%. Pre- to post-drop Schirmer's test scores at Day 1 will be the primary outcome. Some studies found the Day 1 mean differences for pre- to post-drop Schirmer's test score was 8.9, and the 28 Day mean differences for pre- to post-drop Schirmer's test score was 10.6 0.58 mm. If one assumes a clinically meaningful difference of 3 units (SD = 0.58; α of 0.05 and power of 80%), a total of 3 subjects will be needed to determine if there is a significant change in pre- to post-drop Schirmer's test scores. SPEED questionnaire at Days 14 and 28 will be the secondary outcomes. SPEED questionnaire scores of 2.2, 5.0, 6.6, and 9.9 corresponded to having asymptomatic, mild, moderate, and severe dry eye symptoms, and as such a 3 unit change will be considered to be a clinically meaningful difference.11 Asiedu et al. found that the typical subject with moderate dry eye has a mean SD SPEED score of 6.6 , which is the target symptoms severity level of this study.11 If one assumes a clinically meaningful difference of 3 units (SD = 4.1; α of 0.05 and power of 80%), a total of 17 subjects will be needed to determine if there is a significant change in SPEED scores at day 14 or 28. Exploratory outcomes include Likert survey questions; thus, the overall sample size will be inflated to 100 participants to help ensure that representative survey responses are obtained from the participants included in this study.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age.
* Have a history of DED for at least the past 6 months.
* Are currently using Xiidra as directed by their eye care provider for ≥1 month.
* Are symptomatic as determined with SPEED (≥7) and have an abnormal Schirmer test score [≥2 to <10 mm/5 min]) at Screening/Baseline. If Shirmer only qualifies for one eye, that will be the study eye. If Shirmer qualifies for both eyes, the right eye will be the study eye.
* Have corrected distance visual acuity of 20/40 or better.
* Willing to discontinue contact lens wear 24 hours prior to screening visit and throughout the study.

Exclusion Criteria:

* Have a systemic health condition that is known to alter tear film physiology (e.g., primary and secondary Sjögren's syndrome).
* Have a history of ocular surgery within the past 12 months.
* Have a history of severe ocular trauma, active ocular infection or inflammation that is not dry eye related.
* Punctal plugs in place for < 3 months and/or Lacrifill in place for > 5 months.
* Have ever used Accutane
* Currently using ocular medications, including topical anti-inflammatory drops, (other than Xiidra) 1 month prior to enrollment
* Any artificial tear use at enrollment must remain consistent throughout the study.
* Are pregnant or breast feeding.
* Have had a physical meibomian gland treatment withing 1 month of enrollment.
* Initiated, discontinued or changed dose of a systemic medication known to cause ocular drying (e.g., antihistamines or tricyclic antidepressants) within 14 days of the screening visit.
* Have a condition or be in a situation, which in the investigator's opinion, may put the participant at significant risk, may confound the results, or may significantly interfere with their study participation.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Change between pre- and post-drop in unanesthetized Schirmer test score on Day 1 | 1 day
  The Schirmer's strip wetting time/quantity will be measured before and after the drop with quicker and more wetting me considered better.

SECONDARY OUTCOMES:
Change in standardized speed scores | 28 days
  The standardized speed scores will be measured to determine change from baseline to 28 days with lower scores being better.
2 week change in standardized speed scores | 14 days
  The standardized speed scores will be measured to determine change from baseline to 14 days with lower scores being better.